CLINICAL TRIAL: NCT06588426
Title: Clinical Readiness Skin Punch Biopsy Sample Collection
Brief Title: Clinical Readiness Skin Punch Biopsy Sample Collections
Status: Recruiting | Type: Observational
Sponsor: HeartWorks, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IPSC-CL-002
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease (CHD); Congenital Heart Defect
Keywords: CHD; Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample will be manufactured into fibroblasts and induced pluripotent stem cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with congenital heart disease

SUMMARY:
This is a clinical readiness skin punch biopsy sample collection study. This will allow to reduce manufacturing time when patients are identified as eligible to receive product under separate interventional treatment protocol.

DETAILED DESCRIPTION:
This is a clinical readiness skin punch biopsy sample collection study. This will allow to reduce manufacturing time when patients are identified as eligible to receive product under separate interventional treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Congenital heart disease
* Likely to qualify for an active clinical trial under IND 28611 in the future

Exclusion Criteria:

* Previous cardiac transplantation
* Unable or unwilling to consent
* HIV diagnosis
* Hepatitis diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Congenital heart disease patients likely to qualify in the future for treatment using iPSC-CL in an approved clinical trial under IND 28611
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Successful manufacture of induced pluripotent stem cells | 12 months
  Outcome measured will be the manufacture of iPSC that meets pre-determined acceptance criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: General trial information — https://www.mayo.edu/research/clinical-trials/cls-20572361